CLINICAL TRIAL: NCT01348178
Title: Retrospective Follow-up Study After Periacetabular Osteotomy in Adults
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: PAO
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Congenital Deformity of Hip Joints
MeSH Terms: interventions — Tacrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- developmental dysplasia of the hip, PAO: All patients who underwent periacetabular osteotomy from 1999-2007 at the University Hospital of Aarhus
  Interventions: Procedure: Follow-up

INTERVENTIONS:
Procedure: Follow-up — Follow-up
  Other Names: Outcome; THA; WOMAC

SUMMARY:
This is a retrospective study assessing pre- and postoperative radiographic indices of hip dysplasia in order to identify factors predicting failure following Periacetabular Osteotomy (PAO).

DETAILED DESCRIPTION:
Even though the PAO is applied worldwide and is the preferred joint preserving treatment some issues remains unclear and controversial. One is the exact indication for surgery and risk factors for early failure of the procedure. The is a retrospective cohort study assessing pre- and postoperative radiographic indices of hip dysplasia in order to identify factors predicting failure following PAO. The minimum duration of follow-up is 2 years. Failure following PAO is defined by a WOMAC pain score > 10 or the insertion of a total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* PAO from 1999-2007

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent PAO from 1999-2007
Sampling Method: Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2010-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Soballe, Prof. D.Msc, Study Chair — Orthopedic Research Unit, Aarhus University Hospital; Charlotte Hartig-Andreasen, MD, Principal Investigator — Orthopedic Research Unit, Aarhus University Hospital